CLINICAL TRIAL: NCT00068458
Title: A Phase II Randomized Study to Assess the Feasibility of Distance Medicine Based Exercise and Dietary Approaches to Prevent Body Composition Change Occurring During Adjuvant Chemotherapy for Early Stage Breast Cancer
Brief Title: Survival TRaining for ENhancing Total Health (STRENGTH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: U10CA081851 (NIH); U10CA081851 (NIH)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2013-04

CONDITIONS: Breast Cancer; Depression; Weight Changes
Keywords: weight changes; depression; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Depression; Body Weight Changes | interventions — Calcium; Exercise; Fruit; Vegetables; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1: calcium diet (Active Comparator): Calcium-Rich Diet (dietary counseling + materials promoting an intake of 1,200 - 2,500 mg/day).
  Interventions: Dietary Supplement: Calcium-Rich Diet
- Arm 2: Exercise + Calcium-Rich Diet (Active Comparator): Exercise + Calcium Rich Diet (dietary counseling + materials promoting strength training and aerobic activity + a calcium intake of 1,200 - 2,500 mg/day).
  Interventions: Other: Arm 2: Exercise + Calcium-Rich Diet
- Exercise + Fruit & Vegetable, Low Fat + Calcium Diet (Active Comparator): Dietary counseling + materials promoting strength training and aerobic activity + a diet that has < 20% of energy coming from fat and intakes of fruits and vegetables of > 5 servings/day + a calcium intake of 1,200 - 2,500 mg/day. 6 month intervention.
  Interventions: Other: Exercise + Fruit & Vegetable, Low Fat + Calcium Diet

INTERVENTIONS:
Dietary Supplement: Calcium-Rich Diet — 1,200 - 2,500 mg/day. 6 month intervention
  Other Names: Calcium
  Arms: Arm 1: calcium diet
Other: Arm 2: Exercise + Calcium-Rich Diet — Dietary counseling + material promoting strength training an aerobic activity + a calcium intake of 1,200 - 2,500 mg/day. 6 month intervention.
  Other Names: Calcium
  Arms: Arm 2: Exercise + Calcium-Rich Diet
Other: Exercise + Fruit & Vegetable, Low Fat + Calcium Diet — 1,200 - 2,500 Calcium intake per day. 6 month intervention period.
  Other Names: Calcium
  Arms: Exercise + Fruit & Vegetable, Low Fat + Calcium Diet

SUMMARY:
RATIONALE: A home-based exercise and/or diet program may improve the quality of life of breast cancer patients by preventing an increase in body fat and weight and a loss of lean body tissue.

PURPOSE: This randomized phase II trial is studying the effectiveness of three home-based diet and/or exercise programs in preventing weight gain and loss of muscle tissue in women who are receiving chemotherapy for stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of exercise alone or combined with a modified diet as home-based interventions to prevent increases in body fat during adjuvant chemotherapy in women with stage I, II, or IIIA breast cancer.
* Compare the efficacy of these regimens, in terms of reducing gains in adipose tissue, reducing losses in absolute amounts of lean body tissue, reducing gains in weight, influencing levels of biomarkers associated with the risk of breast cancer and/or other comorbid conditions, improving self-efficacy for exercise behaviors, reducing depression, and improving quality of life in these patients.
* Compare the adherence rates to these regimens in these patients.
* Determine the associations between study condition and adherence and change in endpoints in patients treated with these regimens.
* Determine the feasibility of conducting home-based exercise and diet studies using the infrastructure of the cooperative group.

OUTLINE: This is a pilot, randomized, multicenter study. Patients are stratified according to body mass index (no more than 25 kg/m^2 vs more than 25 kg/m^2), race (white vs non-white), and prior exercise history (vigorous exercise of at least 30 minutes, 3 times a week prior to diagnosis) (yes vs no). Patients are randomized to 1 of 3 treatment arms.

* Arm I (calcium-rich diet): Patients receive materials and counseling to promote a diet that contains ample amounts of calcium (1,200-2,500 mg/day).
* Arm II (calcium-rich diet and exercise): Patients receive materials and counseling as in arm I and instruction and materials to promote strength training and endurance exercises.
* Arm III (calcium-rich, high fruit and vegetable, low-fat diet and exercise): Patients receive materials and counseling as in arm II and materials and counseling to consume at least 5 servings of vegetables and fruit per day and limit fat intake to less than 20% of total calories.

In all arms, patients continue regimens for 6 months.

Measurements of body composition, weight, waist circumference, serum levels of insulin, insulin-like growth factor, sex hormone-binding globulin, and total cholesterol are obtained at baseline and 6 months.

Quality of life, depression, diet composition, and physical activity are assessed at baseline and at 3 and 6 months.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 90 patients (30 per treatment arm) will be accrued for this study within 16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Stage I, II, or IIIA
* Scheduled to receive adjuvant chemotherapy OR received 1 prior course of chemotherapy
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal Status

* Premenopausal, defined as at least 1 of the following:

  * Less than 4 months since last menstrual period at diagnosis
  * Follicle-stimulating hormone level in the premenopausal range

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* No calcium-based kidney stones

Cardiovascular

* No angina within the past 6 months
* No myocardial infarction within the past 6 months
* No abnormal MUGA and/or stress test

Other

* Not pregnant or nursing
* Access to a telephone
* Able to read and speak English
* No other prior or concurrent malignancy except curatively treated carcinoma in situ of the cervix or nonmelanoma skin cancer
* No history of hyperthyroidism or hypothyroidism
* No paralysis
* No osteoarthritis with uncontrolled joint pain that would preclude exercise
* No diverticulitis
* No serious medical or psychiatric illness that would preclude giving informed consent or completing study therapy or quality of life questionnaires
* No medical condition that would interfere with body composition assessment
* No medical condition for which unsupervised exercise is contraindicated
* No medical condition for which a high vegetable and fruit diet or a calcium-rich diet is contraindicated

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior bilateral oophorectomy
* No prior amputation
* No concurrent transverse rectus abdominis myocutaneous surgery
* No concurrent surgery

Other

* No concurrent blood-thinners (e.g., coumadin or warfarin)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-09; Primary Completion 2004-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Distance Medicine Based Diet Exercise Program Within the Cooperative Group Setting | 6 months
  Assess estimates of effect sizes and to ascertain potential feasibility of implementing a distance-medicine based diet-exercise program within the cooperative group setting.

CONTACTS AND LOCATIONS:
Overall Officials: Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences; Wendy Demark-Wahnefried, PhD, Principal Investigator — Duke Cancer Institute; Roger T. Anderson, PhD, Study Chair — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina

REFERENCES:
- [Result] Demark-Wahnefried W, Case LD, Blackwell K, Marcom PK, Kraus W, Aziz N, Snyder DC, Giguere JK, Shaw E. Results of a diet/exercise feasibility trial to prevent adverse body composition change in breast cancer patients on adjuvant chemotherapy. Clin Breast Cancer. 2008 Feb;8(1):70-9. doi: 10.3816/CBC.2008.n.005. PMID 18501061